CLINICAL TRIAL: NCT00802139
Title: A Prospective, Randomized, Multi-centered Trial to Compare the Efficacy and Safety of Intravenous Iron Sucrose (Venoferrum®) With Oral Iron Acetyl-transferrin Hydroglycerin (Bolgre®) in Pregnant Women With Iron Deficiency Anemia
Brief Title: Efficacy and Safety Study of Iron Sucrose and Oral Iron Acetyl-transferrin Hydroglycerin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP-VNF-402
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia; pregnant women with iron deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- venoferrum group (Experimental)
  Interventions: Drug: venoferrum(iron sucrose)
- Bolgre group (Active Comparator)
  Interventions: Drug: Bolgre (Iron acetyl-transferase)

INTERVENTIONS:
Drug: venoferrum(iron sucrose) — administer once weekly calculated quantity of Venoferrum® ampoules according to body weight and Hb level.
  Arms: venoferrum group
Drug: Bolgre (Iron acetyl-transferase) — Twice daily administration with Bolgre® soln (one pouch per dosing which is equivalent to 40mg of iron) for 5 weeks
  Arms: Bolgre group

SUMMARY:
multi-center, prospective, randomized, open-labeled, active-drug-controlled, two-parallel-group-comparison(venoferrun group vs Bolgre group)study

ELIGIBILITY:
Inclusion Criteria:

* 30~32nd weeks pregnant women aged over 18 years
* Women who have Hb level of more than 10.0g/dL a week before study initiation
* Patients who agree to participate in this study in writing

Exclusion Criteria:

* Patients who have participated in another clinical study in recent 3 months
* Patients who are prone to acute hemorrhage during pregnancy
* Patients who have shown intolerance to iron therapy
* Hemolytic anemia, hemoglobinopathies (thalassemia, sickle cell)
* Bleeding tendency, hypersplenism
* Chronic heart failure, Class II-IV heart disease, uncontrolled arterial hypertension (DBP ≥ 115mmHg), deep vein thrombosis, thrombocytosis, chronic renal disease
* Severe renal failure patients (2.5 times or more higher plasma creatinine level than high limit of normal state)
* Patients with severe liver dysfunction (2.5 times or more higher AST or ALT than high limit of normal state)
* Patients with doubled or more CK level than high limit of normal state
* Patients who are regarded as ineligible for this study by investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change of plasma hemoglobin level | 5 week

SECONDARY OUTCOMES:
Target Hb achievement rate(11g/dL), Transferrin saturation(%), Ferritin(ng/mL), TIBC(ug/dL), MCV(fl), MCH(pg) and change in reticulocyte counts | 5 week

CONTACTS AND LOCATIONS:
Overall Officials: Kim AM, ph.D, Principal Investigator — Asan hospital OB/Gyn unit
Locations (3):
- South Korea (3):
  - Chonnam National Universitiy Hospital, Kwangju
  - Asan Hospital, Seoul
  - Catholic University of Korea Kangnam St. Mary's Hospital, Seoul